CLINICAL TRIAL: NCT01487252
Title: Circadian Phase Assessments at Home
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Rush University Medical Center (Other)
Collaborators: National Center for Complementary and Integrative Health (NCCIH) (NIH)
Responsible Party: Principal Investigator, Helen Burgess, Professor, Rush University Medical Center
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Diagnostic
Other Study IDs: AT007104
Record Dates: First submitted 2011-12-02; First posted 2011-12-07 (Estimated); Last update posted 2017-04-12 (Actual); Status verified 2017-04

CONDITIONS: Healthy Controls; Delayed Sleep Phase

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Healthy Controls (Active Comparator)
  Interventions: Behavioral: At home saliva sampling
- Delayed Sleep Phase Disorder (Active Comparator)
  Interventions: Behavioral: At home saliva sampling

INTERVENTIONS:
Behavioral: At home saliva sampling — Saliva samples taken every half an hour in evening before bedtime.

SUMMARY:
An estimated 23 million Americans, including adolescents and the elderly, suffer from circadian rhythm sleep disorders, such as delayed sleep phase disorder, advanced sleep phase disorder and winter depression. These conditions are characterized by persistent insomnia and/or excessive daytime sleepiness, impaired performance, reduced well being and lower quality of life. The negative symptoms result from a misalignment between the timing of sleep and the internal circadian clock. Clinical research has demonstrated that circadian rhythm sleep disorders are most effectively diagnosed (differentiated from other causes of insomnia) and treated if each individual patient's circadian phase is known. The timing of the master internal circadian clock is most reliably measured from the onset of the endogenous circadian rhythm of melatonin, a neuroendocrine hormone, as measured in dim light (dim light melatonin onset, or "DLMO"). However to date the reliable and valid assessment of the DLMO is limited to the research laboratory setting.

This study is to test a streamlined procedure for the accurate assessment of circadian phase (DLMO) outside of the laboratory that will provide clinicians and researchers with a novel diagnostic and research tool. In this way the underlying neurobiological cause of a patient's insomnia and/or circadian rhythm disorder can more readily be diagnosed and treated.

Specific Aim 1 is to validate procedures for at-home circadian phase assessment in a sample of healthy people. Validation will occur by (1) objectively measuring compliance to the at-home procedures and (2) comparing DLMOs collected at home to DLMOs collected in the laboratory, in a within-subjects counterbalanced design. Specific Aim 2 is to validate the same at home procedures in patients with delayed sleep phase disorder. Specific Aim 3 is to conduct rigorous analyses to inform future users which subject characteristics and light levels predict (1) compliance to the at home procedures and (2) valid at-home DLMOs.

The results of this 3 year study will have substantial implications for the translation of basic and clinical research to the community: (1) the diagnosis and treatment of insomnia and circadian rhythm sleep disorders will be significantly enhanced, thus improving public health and safety, mood and quality of life, (2) community participation in research will be improved, particularly in vulnerable and under represented populations, thus increasing scientific knowledge and (3) research and clinical costs will be substantially reduced.

ELIGIBILITY:
Inclusion Criteria:

* Healthy adult volunteers or people with Delayed Sleep Phase Disorder

Exclusion Criteria:

* Color blindness with the Ishihara test

Ages: 18 Years to 69 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 73 (Actual)
Dates: Start 2011-12; Primary Completion 2014-12 (Actual); Study Completion 2015-05 (Actual)

PRIMARY OUTCOMES:
Dim Light Melatonin Onset | 9 days
  The DLMO is assessed twice at home and twice in the laboratory.

CONTACTS AND LOCATIONS:
Locations (1):
- Rush University Medical Center, Chicago, Illinois, United States

REFERENCES:
- [Derived] Burgess HJ, Park M, Wyatt JK, Rizvydeen M, Fogg LF. Sleep and circadian variability in people with delayed sleep-wake phase disorder versus healthy controls. Sleep Med. 2017 Jun;34:33-39. doi: 10.1016/j.sleep.2017.02.019. Epub 2017 Mar 14. PMID 28522096
- [Derived] Burgess HJ, Park M, Wyatt JK, Fogg LF. Home dim light melatonin onsets with measures of compliance in delayed sleep phase disorder. J Sleep Res. 2016 Jun;25(3):314-7. doi: 10.1111/jsr.12384. Epub 2016 Feb 5. PMID 26847016
- [Derived] Burgess HJ, Wyatt JK, Park M, Fogg LF. Home Circadian Phase Assessments with Measures of Compliance Yield Accurate Dim Light Melatonin Onsets. Sleep. 2015 Jun 1;38(6):889-97. doi: 10.5665/sleep.4734. PMID 25409110